CLINICAL TRIAL: NCT00031733
Title: A Phase II Randomized Trial of a Vaccine Combining Tyrosinase/GP100/MART-1 Peptides Emulsified With Montanide ISA 51 With Interleukin-12 With Alum or GM-CSF for Patients With Resected Stages IIB/C, III and IV Melanoma
Brief Title: Vaccine Therapy and Interleukin-12 With Either Alum or Sargramostim After Surgery in Treating Patients With Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000069220 (10M-01-1); LAC-USC-10M011; LAC-USC-IRB-013030; NCI-5506
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: iris melanoma; ciliary body and choroid melanoma, small size; ciliary body and choroid melanoma, medium/large size; extraocular extension melanoma; recurrent intraocular melanoma; stage II melanoma; stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — MART-1 Antigen; incomplete Freund's adjuvant; Interleukin-12 Subunit p35; sargramostim; Aluminum Hydroxide; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: MART-1 antigen
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant
Biological: recombinant interleukin-12
Biological: sargramostim
Biological: tyrosinase peptide
Drug: alum adjuvant
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Vaccines made from peptides may make the body build an immune response. Combining vaccine therapy with interleukin-12 and either alum or sargramostim may kill more tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of combining vaccine therapy with interleukin-12 and either alum or sargramostim in treating patients who have undergone surgery for stage II, stage III, or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the immune reactivity in patients with resected stage IIB, IIC, III, or IV melanoma vaccinated with tyrosinase, gp100, and MART-1 peptides emulsified with Montanide ISA-51 with interleukin-12 and either alum adjuvant or sargramostim (GM-CSF).

OUTLINE: This is a randomized study. Patients are stratified according to disease stage (cutaneous stage IIB, IIC, III, and IV vs ocular and mucosal stage III and IV). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive vaccine with tyrosinase:368-376 (370D)/gp100:209-217 (210M)/MART-1:26-27 (27L) peptides emulsified with Montanide ISA-51 (ISA-51), low-dose interleukin-12 (IL-12) subcutaneously (SC), and alum adjuvant SC on day 1 of weeks 1, 3, 5, 7, 11, 15, 19, 27, and 53.
* Arm II: Patients receive peptide vaccine emulsified with ISA-51, high-dose IL-12 SC, and alum adjuvant SC on day 1 of weeks 1, 3, 5, 7, 11, 15, 19, 27, and 53.
* Arm III: Patients receive peptide vaccine emulsified with ISA-51 on day 1 and low-dose IL-12 SC and sargramostim (GM-CSF) SC on days 1-5 of weeks 1, 3, 5, 7, 11, 15, 19, 27, and 53.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 60 patients (20 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage IIB, IIC, III, or IV cutaneous melanoma OR stage III or IV ocular or mucosal melanoma

  * Resected or rendered disease-free
* HLA-A2.1-positive by standard cytotoxicity assay
* Tumor tissue must be available for analysis of gp100 staining and tyrosinase and MART-1 expression by immunohistochemistry

  * Must be positive for at least 1 antigen
* Failed, ineligible for, or refused prior interferon alfa

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL
* No bleeding disorder

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGOT/SGPT no greater than 2.5 times normal
* No coagulation disorder
* Hepatitis surface antigen B negative
* Hepatitis C negative

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No major cardiovascular illness

Pulmonary:

* No major respiratory illness

Immunologic:

* No prior uveitis
* No prior autoimmune inflammatory eye disease
* No immune hemolytic anemia
* No other active autoimmune disease

Other:

* HIV negative
* No major gastrointestinal illness
* No other malignancy within the past 5 years except squamous cell skin cancer or carcinoma in situ of the cervix curatively treated at least 30 days ago
* No major systemic infection (e.g., pneumonia or sepsis)
* No other major medical illness
* No prior allergic reaction to Montanide ISA-51 or alum adjuvant
* No requirement for steroid therapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No prior tyrosinase:368-376 (370D), gp100:209-217 (210M), or MART-1:26-35 (27L) peptides

Chemotherapy:

* At least 1 month since prior adjuvant chemotherapy for this disease
* No concurrent adjuvant chemotherapy

Endocrine therapy:

* No concurrent steroids

Radiotherapy:

* At least 1 month since prior radiotherapy for this disease
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* At least 1 month since other prior therapy, including adjuvant therapy, for this disease
* No other concurrent therapy, including adjuvant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-02; Primary Completion 2004-12 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Weber, MD, PhD, Study Chair — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California, United States